CLINICAL TRIAL: NCT06996548
Title: Investigation of the Relationship Between Sarcopenia and Paclitaxel-Induced Neuropathy in Early Stage Breast Cancer Patients (Neuro-Sarc)
Brief Title: Sarcopenia and Paclitaxel-Induced Neuropathy in Early Stage Breast Cancer (Neuro-Sarc)
Acronym: Neuro-Sarc
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, Principal Investigator, Specialist in Medical Oncology, Department of Medical Oncology, Gazi University
Other Study IDs: NEURO-SARC-001; 2024-10/157 (Other: Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia; Paclitaxel Induced Neuropathy; Breast Carcinoma
Keywords: Paclitaxel; Breast cancer; Sarcopenia; Neuropathy
MeSH Terms: conditions — Sarcopenia; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paclitaxel-Treated Early Stage Breast Cancer Patients: Patients aged 18 years or older with early-stage breast cancer who received neoadjuvant or adjuvant paclitaxel-based chemotherapy, including paclitaxel plus carboplatin or paclitaxel plus trastuzumab/pertuzumab. Neuropathy was assessed before and after chemotherapy, and skeletal muscle index was measured from baseline CT scans.

SUMMARY:
This prospective observational study aims to investigate the relationship between sarcopenia and the development of paclitaxel-induced peripheral neuropathy in patients with early-stage breast cancer. The study was conducted between November 1, 2024, and May 6, 2025, across three oncology centers in Turkey. Skeletal muscle index (SMI) was calculated using pre-treatment computed tomography (CT) scans at the third lumbar vertebra (L3) level. Neuropathy assessment was performed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20-item scale (EORTC QLQ-CIPN20) before and after paclitaxel treatment. Patients reporting neuropathy symptoms were referred for electromyography (EMG) to confirm diagnosis, and neuropathy was graded according to the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0). The association between baseline sarcopenia and both the incidence and severity of neuropathy was analyzed. The findings may help identify patients at higher risk of neurotoxicity from paclitaxel-based chemotherapy.

DETAILED DESCRIPTION:
This multicenter prospective observational study was designed to evaluate whether baseline sarcopenia is associated with the development and severity of peripheral neuropathy in patients receiving paclitaxel as part of neoadjuvant or adjuvant chemotherapy for early-stage breast cancer.

Patients aged 18 years or older with histologically confirmed early-stage breast cancer who received paclitaxel-based treatment (including combinations with carboplatin, trastuzumab, or pertuzumab) were included. Skeletal muscle index (SMI) was calculated from computed tomography (CT) scans at the third lumbar vertebra (L3) level, taken prior to paclitaxel initiation.

Neuropathy was assessed at baseline and after the final paclitaxel cycle using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20-item scale (EORTC QLQ-CIPN20). Patients with symptoms suggestive of neuropathy were referred for electromyography (EMG) confirmation, and neuropathy severity was classified according to the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).

The primary aim was to evaluate the association between sarcopenia and the occurrence of chemotherapy-induced peripheral neuropathy (CIPN). Secondary outcomes included the relationship between sarcopenia and the severity grade of neuropathy.

This study seeks to provide insights into risk stratification for CIPN and guide supportive care strategies in early-stage breast cancer patients undergoing taxane-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed early-stage breast cancer
* Planned to receive neoadjuvant or adjuvant paclitaxel-based chemotherapy
* Patients receiving paclitaxel-carboplatin or paclitaxel-trastuzumab-pertuzumab regimens are also eligible
* Provided written informed consent

Exclusion Criteria:

* Age < 18 years
* No pathological diagnosis of breast cancer
* Refusal to participate in the study
* Male patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as women and have a biologically female sex assigned at birth are eligible to participate in this study due to the focus on early-stage breast cancer.
Study Population: The study population consisted of adult female patients diagnosed with early-stage breast cancer and treated with neoadjuvant or adjuvant paclitaxel-based chemotherapy regimens at three oncology centers in Turkey. Patients were enrolled consecutively if they met the inclusion criteria and provided informed consent. Data were collected prospectively, including pre-treatment CT scans for muscle mass analysis and neuropathy assessments.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Paclitaxel-Induced Peripheral Neuropathy | From baseline to end of paclitaxel treatment (approximately 12 weeks)
  The proportion of patients developing chemotherapy-induced peripheral neuropathy (CIPN) during or after paclitaxel treatment. Neuropathy will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20-item scale (EORTC QLQ-CIPN20; score range: 0 to 100, where higher scores indicate worse symptoms). Electromyography (EMG) will be used to confirm clinical diagnosis when needed.

SECONDARY OUTCOMES:
Severity of Chemotherapy-Induced Peripheral Neuropathy | At the end of paclitaxel treatment (approximately 12 weeks)
  Neuropathy severity will be graded using the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0), ranging from Grade 1 (mild) to Grade 4 (disabling). The correlation between baseline sarcopenia status and the highest grade of neuropathy observed will be evaluated.
Association Between Sarcopenia and Peripheral Neuropathy | From baseline to end of treatment (approximately 12 weeks)
  The study will evaluate whether sarcopenia (defined by skeletal muscle index [SMI] measured on pre-treatment computed tomography [CT] scans) is correlated with the incidence and severity of paclitaxel-induced peripheral neuropathy (CIPN), as determined by EORTC QLQ-CIPN20 scores and CTCAE v4.0 grades.

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Deliktas, MD, Principal Investigator — Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Locations (3):
- Turkey (Türkiye) (3):
  - Ankara Etlik City Hospital, Ankara, Yenimahalle
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara, Yenimahalle
  - Gazi University, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies and the absence of a data sharing infrastructure. The study involves sensitive clinical information, and no formal mechanism for anonymized data sharing is currently in place.

REFERENCES:
- [Result] Onur ID, Ozdemir PA, Akdogan O, Baskurt K, Kara MI, Kalkan DO, Uyar GC, Sutcuoglu O, Oksuzoglu B, Gurler F, Savran B, Ciledag N, Ates O, Yildiz F. Impact of sarcopenia on paclitaxel-induced peripheral neuropathy in early-stage breast cancer: a prospective observational study (the neuro-sarc study). Support Care Cancer. 2025 Nov 14;33(12):1061. doi: 10.1007/s00520-025-10157-w. PMID 41238950